CLINICAL TRIAL: NCT04301388
Title: A Comparison of the Effectiveness in Management of Threatened Preterm Labor Between Cervical Length-based Approach and Conventional Approach: A Randomized Control Trial
Brief Title: Management of Threatened Preterm Labor by Cervical Length-based Approach or Conventional Approach
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We unable to include the participants as we expected. Only 1 case included after 4 months of recruitment so we decided to withdrawn the study. This is because of COVID-19 pandemic, result in decreasing in the number of patient visiting our insitute.
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Kuntharee Traisrisilp, Assistant professor, Chiang Mai University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OBG-2562-06699
Record Dates: First submitted 2020-03-06; First posted 2020-03-10 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Preterm Delivery Within 7 Day After Admission

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TVCL-based (Experimental): Monitor progression of labor by shortening of cervix examined by transvaginal cervical length
  Interventions: Procedure: Transvaginal ultrasound
- Conventional-based (Active Comparator): Monitor progression of labor by per vaginal exam to detect cervical change
  Interventions: Procedure: Transvaginal ultrasound

INTERVENTIONS:
Procedure: Transvaginal ultrasound — Transvaginal ultrasound to measure cervical length if persist regular uterine contraction

SUMMARY:
To compare the effectiveness of treatment of threatened preterm labor between transvaginal cervical length-based approach and conventional approach (Per vaginal examination)

ELIGIBILITY:
Inclusion Criteria:

* Pregnant with symptoms of threatened preterm labor which refer to regular uterine contractions at least 1 time in every 10 minutes and persist for 30 minute without cervical dilatation or cervical dilation ≤ 1 cm and < 80% of effacement.
* Age ≥ 18 years
* Singleton pregnancy
* 24 0/7 - 33 6/7 weeks of gestation
* Uneventful antenatal care or low-risk pregnancies

Exclusion Criteria:

* The definitive diagnosis of true labor
* Proceed to the active phase of labor
* Age < 18 years
* Multiple pregnancies
* < 24 or ≥ 34 weeks of gestation
* Fetal chromosomal or structural abnormalities
* Abnormal fetal growth
* Abnormal amniotic fluid
* Evidence of placenta previa
* Significant vaginal bleeding that cannot be ruled out placenta previa
* Evidence of rupture of membranes
* Evidence of intrauterine infection
* Evidence of uterine malformation
* Evidence of lethal fetal malformation
* Unable to communicate or understand the information of the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Study in pregnant women
Enrollment: 0 (Actual)
Dates: Start 2020-01-22 (Actual); Primary Completion 2020-05-04 (Actual); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Number of cases with delivery within 7 day after admission | From admission to no uterine contraction in 10 minute
  In case of threatened preterm labor if detection the progression of labor by transvaginal cervical length, the rate of delivery within 7 days will less or more than conventional group.

SECONDARY OUTCOMES:
The number of tocolysis courses, length of hospital stay | From admission to no uterine contraction in 10 minute
  In case of tocolytic used for stop labor. The number of medication will be recorded.
The number of steroid courses | From admission to no uterine contraction in 10 minute
  In case of stop labor, the course of steroid for promote lung maturity is recorded.

CONTACTS AND LOCATIONS:
Locations (2):
- Thailand (2):
  - Kuntharee Traisrisilp, Chiang Mai
  - Maharaj Nakorn ChiangMai Hospital, Chiang Mai

IPD SHARING:
Plan to Share IPD: No